CLINICAL TRIAL: NCT03292887
Title: Hunter Outcome Survey: A Global, Multi-Center, Long-Term, Observational Registry of Patients With Hunter Syndrome (Mucopolysaccharidosis Type II, MPS II)
Brief Title: Hunter Outcome Survey (HOS)
Acronym: HOS
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HOS
Record Dates: First submitted 2017-09-18; First posted 2017-09-26 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hunter Syndrome
Keywords: Mucopolysaccharidosis II; Hunter Syndrome; Enzyme Replacement Therapy; Lysosomal; Glycosaminoglycans
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elaprase Treated: Participants with Hunters Syndrome received or receiving treatment with Elaprase as prescribed by their physician following locally approved prescribing information.
- Elaprase Non-Treated: Participants received no treatment for Hunters Syndrome.

SUMMARY:
The purpose of this study is to collect data that will increase understanding of Hunter syndrome. The data from HOS may provide guidance to healthcare professionals about disease treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Hunter syndrome (biochemically and/or genetically)
2. Signed and dated written informed consent, as per either a or b below:

   1. Prospective Participants: Signed and dated written informed consent from the participant or, for participants aged less than (<) 18 years (<16 years in Scotland), parent and/or participant's legally authorized representative (LAR), and assent of the minor where applicable.

      informed consent must be obtained from LARs for cognitively impaired participants, where applicable.

      OR
   2. Historical Participants: Signed and dated informed consent from the participant's LAR (where allowed by relevant individual country or site regulations/laws). .

Exclusion Criteria:

1. Participants enrolled in an interventional clinical trial are not eligible. Participants may re-enroll once they have completed or withdrawn from the other clinical study.
2. Participants receiving treatment for Hunter syndrome with an ERT product other than Elaprase are not eligible. Participants may enroll or re-enroll once they have stopped treatment with another ERT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The HOS registry is open to all participants (both alive and deceased) with Hunter syndrome who are untreated or who are receiving/received treatment with Elaprase, including participants who are alive at HOS enrollment (referred to as "Prospective Patients") and participants who are deceased at HOS enrollment (referred to as "Historical Patients").
Sampling Method: Non-Probability Sample
Enrollment: 1443 (Actual)
Dates: Start 2005-10-03 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Infusion-related Reactions (IRRs) | Baseline to year 17
  An Infusion-related reaction (IRR) is an adverse event (AE) that occurs during or within 24 hours of an infusion and with evidence of a causal relationship with Elaprase.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to year 17
  An AE is any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in the registry, whether or not considered product-related. This includes an exacerbation of a pre-existing condition. An AE or adverse drug reaction (ADR) that meets one or more of the following criteria/outcomes is classified as serious whether considered to be related to the pharmaceutical product or not: death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalizations, a persistent or significant disability or incapacity, a congenital anomaly or birth defect and important medical events.
Number of Participants With Positive Antibody Response | Baseline to year 17
  Immunogenicity is determined by time to first positive antibody response (antibody level and isotype), antibody titer, isotype, and neutralizing antibodies.
Change in Urinary Glycosaminoglycan (GAG) Levels | Baseline to year 17
  Change in urinary GAG levels from the start of ERT is reported.
Change in Height | Baseline to year 17
  Change in height from the start of ERT will be reported.
Change in Weight | Baseline to year 17
  Change in weight from the start of ERT will be reported.
Change in Head Circumference and Corresponding Calculated Z-scores | Baseline to year 17
  Change in head circumference with the corresponding Z-scores from the start of ERT will be reported.
Change in Distance Walked in the 6-minute Walk Test | Baseline to year 17
  Change in distance walked in 6-minute walk test from the start of ERT is reported.
Left Ventricular Mass Index (LVMI) | Baseline to year 17
  Change in LVMI will be assessed as calculated by echocardiography.
Change in Forced Expiratory Volume in 1 Second (FEV1) | Baseline to year 17
  Change in pulmonary function from the start of ERT will be reported as measured by forced expiratory volume in 1 second (FEV1).
Change in Forced Vital Capacity (FVC) | Baseline to year 17
  Change in pulmonary function from the start of ERT will be reported as measured by forced vital capacity (FVC).
Change in Liver and Spleen Size | Baseline to year 17
  Change in liver and spleen size as estimated by palpation will be reported.
Prevalence of Cardiac and Pulmonary-related Hospitalizations | Baseline to year 17
  Prevalence of cardiac and pulmonary-related hospitalizations will be reported.
Age at the Time of Death | Baseline to year 17
  Age at the time of death will be reported.
Cause of Death | Baseline to year 17
  Causes of death will be reported

SECONDARY OUTCOMES:
Natural History of Untreated Participants With Hunter Syndrome | Baseline to year 17
  Evaluation of signs and symptoms for the natural history of disease: hepatosplenomegaly, central nervous system involvement, skeletal involvement, ear, nose, and throat signs and symptoms, pulmonary signs and symptoms and cardiac signs and symptoms will be reported.
Dosing Regimens of Elaprase for Prescribed Dose in Participants With Hunter Syndrome | Baseline to year 17
  Dosing regiments of Elaprase will be evaluated for prescribed dose.
Dosing Regimens of Elaprase for Administered Dose in Participants With Hunter Syndrome | Baseline to year 17
  Dosing regiments of Elaprase will be evaluated for administered dose.
Dosing Regimens of Elaprase for Total Infusion Time in Participants With Hunter Syndrome | Baseline to year 17
  Dosing regiments of Elaprase will be evaluated for total infusion time.
Dosing Regimens of Elaprase for Missed Infusions in Participants With Hunter Syndrome | Baseline to year 17
  Dosing regiments of Elaprase will be evaluated for missed infusions.
Dosing Regimens of Elaprase for Reason for Missed Infusions. | Baseline to year 17
  Dosing regiments of Elaprase will be evaluated for reason for missed infusions.
Assessment of Hunter Syndrome on Health-related Quality of Life (HRQL) Using Hunter Syndrome-Functional Outcomes for Clinical Understanding Scale (HS-FOCUS) | Baseline to year 17
  HS-FOCUS was developed as disease-specific measure of the impact of Hunter syndrome on HRQL. The HS-FOCUS is designed to gather information on the participant's daily life and wellbeing, satisfaction with treatment, and hospitalizations, as well as on how Hunter syndrome impacts participant's general quality of life. HS-FOCUS includes 2 validated components: a parent version and a patient self-reported version for those over age 12 years. The HS-FOCUS Version 2.0 contains 6 functional status domains: Walking/Standing, Reach/Grip, Sleeping, Schooling/Work, Activities, and Breathing. Items are scored using a response scale from 0 to 4, with ="0" expressing being able to complete the activity-related functions "without any difficulty" and "4" as "unable to do so. Scores are averaged to calculate the 6 function domain scores and the Overall Function Score, with higher scores corresponding to a higher degree of incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Shire, Lexington, Massachusetts, United States

REFERENCES:
- [Derived] Muenzer J, Amartino H, Giugliani R, Harmatz P, Lin SP, Link B, Molter D, Ramaswami U, Scarpa M, Botha J, Audi J, Burton BK. Unmet needs of adults living with mucopolysaccharidosis II: data from the Hunter Outcome Survey. Orphanet J Rare Dis. 2025 Jul 1;20(1):319. doi: 10.1186/s13023-024-03464-8. PMID 40598289
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fcf4db2bf003ab46821